CLINICAL TRIAL: NCT07192081
Title: Comparative Efficacy of Intravenous Labetalol and Lignocaine in Mitigating Hemodynamic Responses to Laryngoscopy During Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Comparative Efficacy of Intravenous Labetalol and Lignocaine in Mitigating Hemodynamic Responses to Laryngoscopy During Laparoscopic Cholecystectomy
Acronym: LAB-LIG RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Waseem Ullah (Other Government)
Collaborators: Hayatabad Medical Complex (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Waseem Ullah, Registrar, Lady Reading Hospital, Pakistan
Organization: Lady Reading Hospital, Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPSP/REU/ANS-2023-021-3099
Record Dates: First submitted 2025-09-15; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Intubation; Anesthesia; Laparoscopic Cholecystectomy; Hemodynamic Response to Laryngoscopy
Keywords: Attenuation of Sympathetic Response; Perioperative Management; Randomized Controlled Trial; Endotracheal Intubation; Hemodynamic Stability; Lignocaine; Labetalol
MeSH Terms: interventions — Labetalol; Lidocaine

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, single-blind, parallel-arm trial comparing IV labetalol and lignocaine in adult patients undergoing laparoscopic cholecystectomy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group allocation. The anesthesiologist administering the intervention will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labetalol Group (Experimental): Patients in this arm will receive intravenous labetalol at a dose of 0.25 mg/kg over 60 seconds, 3 minutes prior to laryngoscopy and intubation.
  Interventions: Drug: Labetalol
- Lignocaine Group (Active Comparator): Patients in this arm will receive intravenous lignocaine at a dose of 1.5 mg/kg over 60 seconds, 3 minutes prior to laryngoscopy and intubation.
  Interventions: Drug: Lignocaine

INTERVENTIONS:
Drug: Labetalol — Labetalol 0.25 mg/kg intravenous bolus over 60 seconds, administered 3 minutes before laryngoscopy.
  Arms: Labetalol Group
Drug: Lignocaine — Lignocaine 1.5 mg/kg intravenous bolus over 60 seconds, administered 3 minutes before laryngoscopy.
  Arms: Lignocaine Group

SUMMARY:
Laryngoscopy and intubation during laparoscopic cholecystectomy often cause sudden increases in heart rate and blood pressure, which can be harmful in some patients. Medications such as labetalol and lignocaine are commonly used to reduce this hemodynamic response. This randomized controlled trial at Hayatabad Medical Complex, Peshawar, will compare intravenous labetalol (0.25 mg/kg) and lignocaine (1.5 mg/kg), administered 3 minutes before laryngoscopy. A total of 116 patients undergoing elective laparoscopic cholecystectomy will be randomly assigned to either drug group. The primary goal is to determine which drug is more effective in keeping heart rate and mean arterial pressure within ±20% of baseline during and after intubation. The study will also record blood pressure trends, intubation details, rescue medications, and adverse events such as bradycardia or hypotension. Results will help guide anesthesiologists in selecting the safer and more effective option to maintain cardiovascular stability during surgery.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the standard surgical treatment for symptomatic gallstones. However, laryngoscopy and endotracheal intubation during anesthesia often trigger a sympathetic surge, resulting in tachycardia and hypertension. These hemodynamic changes, although short-lived, may increase perioperative risk, especially in patients with limited cardiovascular reserve.

Labetalol, a combined α1- and β-adrenergic antagonist, reduces both heart rate and arterial pressure by blunting sympathetic activity. Lignocaine, an amide local anesthetic, also exhibits sympatholytic effects when given intravenously. Both agents are widely used in anesthesia practice, but direct head-to-head evidence in the setting of laparoscopic cholecystectomy remains limited.

This randomized controlled study will evaluate and compare the efficacy of intravenous labetalol and lignocaine in attenuating pressor and tachycardic responses to laryngoscopy. The trial will include adult ASA I patients scheduled for elective laparoscopic cholecystectomy. Participants will be randomly assigned to receive either labetalol 0.25 mg/kg or lignocaine 1.5 mg/kg intravenously, 3 minutes before laryngoscopy. Hemodynamic variables (heart rate, systolic, diastolic, and mean arterial pressures) will be tracked peri-intubation. The occurrence of adverse events such as bradycardia, hypotension, or allergic reactions will also be monitored.

By directly comparing these two commonly used drugs in a controlled setting, the study aims to clarify which provides superior cardiovascular stability during airway instrumentation. Findings will contribute to evidence-based guidance for anesthesiologists in selecting pharmacologic strategies that minimize perioperative risk in laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA Grade I and II
* Age 18 to 60 years
* Elective laparoscopic cholecystectomy
* Both genders
* Informed consent given

Exclusion Criteria:

* Hypersensitivity to labetalol/lignocaine
* Hypertensive on antihypertensives
* ASA Grade III or more
* Cardiovascular, renal, hepatic, or endocrine issues
* Pregnant/lactating
* BMI ≥ 35
* Anticipated difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-01-04 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) Following Laryngoscopy | From 5 minutes before induction to 10 minutes after intubation.
  To evaluate and compare the effect of intravenous labetalol and lignocaine on systolic blood pressure changes in response to laryngoscopy during induction for laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure (DBP) | From 5 minutes before induction to 10 minutes after intubation.
  To assess diastolic blood pressure response post-laryngoscopy between both groups.
Change in Mean Arterial Pressure (MAP) | From 5 minutes before induction to 10 minutes after intubation..
  To compare MAP variations post-induction and post-laryngoscopy.
Change in Heart Rate | From 5 minutes before induction to 10 minutes after intubation.
  To evaluate the impact of interventions on HR response to laryngoscopy.
Incidence of Adverse Events | From induction through recovery (approx. 1 hour)
  Number of participants experiencing side effects such as bradycardia, hypotension, or allergic reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayatabad Med Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to institutional policies, privacy concerns, and limitations in data-sharing infrastructure.